CLINICAL TRIAL: NCT06249789
Title: Enhancing Recovery in Hip Fracture Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Principal Investigator, Haleh Saadat, Associate Clinical Professor of Anesthesiology, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HHC-2023-0269.
Record Dates: First submitted 2024-01-25; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Intervention Model Description: Research Design & Procedures: Patients will be categorized into two groups:
  Arm A (spinal anesthesia):
  Patients will receive an ultrasound-guided Fascia Iliaca Compartment Block (FICB) injection.
  A single-shot spinal anesthetic will be administered. Propofol will be used for intraoperative sedation, ensuring patient responsiveness.
  Fentanyl will be given as needed for pain relief.
  Arm B (general anesthesia):
  Patients will receive an ultrasound-guided Fascia Iliaca Compartment Block (FICB) injection.
  A general anesthetic will be administered using appropriate airway management devices, with Propofol infusion for maintenance.
Who Masked: Outcomes Assessor
Masking Description: The outcome evaluators and analysts would be unaware of which treatment the participants received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Spinal Anesthesia (Active Comparator): This arm gets preoperative single-dose spinal anesthesia plus an ultrasound-guided Fascia Iliaca Compartment Block (FICB).
  Interventions: Procedure: Spinal Anesthesia
- General Anesthesia (Active Comparator): This arm gets preoperative general anesthesia plus an ultrasound-guided Fascia Iliaca Compartment Block (FICB).
  Interventions: Procedure: General Anesthesia

INTERVENTIONS:
Procedure: Spinal Anesthesia — Participants in this arm will receive single-shot spinal anesthesia with 12-15 mg of either 0.05% or 0.75% bupivacaine (iso or hyperbaric) once before surgery. Additionally, they will undergo an ultrasound-guided nerve block called the Fascia Iliaca Compartment Block (FICB ) in combination with spinal anesthesia.
  Arms: Spinal Anesthesia
Procedure: General Anesthesia — Participants in this group will be given a combination of general anesthesia and a nerve block. General anesthesia involves the use of a sedative called propofol, along with devices to ensure that the airway remains open during the procedure. Additionally, they will undergo an ultrasound-guided nerve block known as the Fascia Iliaca Compartment Block (FICB) in combination with spinal anesthesia.
  Arms: General Anesthesia

SUMMARY:
The purpose of this study is to look at how two different types of anesthesia, spinal and general, affect participants with broken hips who are getting a special kind of pain block before surgery.

Researchers will check:

* How quickly patients are ready for anesthesia
* How long they stay in the recovery room after surgery
* How much pain medicine they need during recovery
* If they experience any confusion
* If one group has complications in one of these anesthesia techniques?

Participants in the study will be put into one of two groups by chance to see if there's a difference in their recovery.

DETAILED DESCRIPTION:
This clinical trial aims to compare two common anesthesia techniques, spinal and general anesthesia, combined with a preoperative nerve block called the Fascia Iliaca Compartment Block (FICB). The objective is to understand how these methods affect patients undergoing hip fracture surgery.

The main questions this study aims to answer are:

* Does the choice between spinal and general anesthesia influence how quickly patients recover from anesthesia?
* Does it affect how long patients stay in the Post-Anesthesia Care Unit (PACU)?
* Does it change the amount of opioid pain medication needed after surgery?
* Do the different anesthesia types impact the occurrence of postoperative delirium?
* Do they affect the length of the hospital stay after surgery?
* Do they lead to different rates of post-operative complications?

Participants will:

* Receive either spinal anesthesia with Fascia Iliaca Compartment Block (FICB) (Arm A) or general anesthesia with Fascia Iliaca Compartment Block (FICB) (Arm B).
* Undergo an ultrasound-guided FICB injection.
* Receive appropriate anesthesia and sedation during surgery.
* Be monitored for pain and provided with pain relief as needed.

The study's broader objectives include enhancing patient safety and satisfaction, reducing hospital readmission rates, lowering healthcare costs, and improving overall healthcare practices. Although direct benefits to participants are not guaranteed, the findings will inform better care for future patients with hip fractures.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting all of the following criteria will be included:

* any gender
* any race/ethnicity
* age 60-89 years
* admitted to St Vincent's Medical Center (SVMC) for elective hip fracture: intramedullary (IM) nailing or open reduction internal fixation (ORIF)
* able to communicate in English or Spanish

Exclusion Criteria:

Patients meeting any of the following criteria will be excluded:

* age <60 or ≥90 years old
* Body Mass Index (BMI) >50 kg/m2
* not ambulatory prior to the fracture
* have a current daily Morphine Equivalent Dose (MED) surpassing 20-milligram equivalents (MME)
* communicate in a language other than English or Spanish (due to lack of availability of translators and issues with patient management if dependent on the Hartford Health Center (HHC) language line)
* history of substance abuse, which might interfere with anesthesia administration, pain management, and overall study outcomes
* have undergone previous hip surgery on the side of the fracture
* refusal to participate or lack of signed study informed consent from the patient or their proxy (in cases where patients lack the capacity to consent)
* have absolute contraindications to spinal anesthesia, determined preoperatively by the regional anesthesiologist in charge, such as:

  * suspected or known coagulopathy (congenital or acquired)
  * current usage of anticoagulant medication within a timeframe deemed inappropriate for neuraxial block by the American Society of Regional Anesthesia guidelines
  * unrepaired critical or severe aortic stenosis
  * active skin infection at the needle insertion site
  * elevated intracranial pressure precluding Dural puncture
* have an increased risk (assessed by reviewing the patient's medical record) for malignant hyperthermia (MH), such as patients with any prior personal or family history of MH or adverse reactions to anesthesia due to MH

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Measuring Pain: Visual Analog Scale (VAS) | Postoperative Anesthesia Unit (PACU) stay: Approximately 2-4 hours from arrival to PACU to release to the floor.
  The pain scale ranges from 0, no pain, to 10, the worst pain imaginable.
Post-anesthesia Care Unit (PACU) Opioid consumption | Approximately 2-4 hours: From the moment the patient arrives in the Post Anesthesia Care Unit (PACU) until their departure to the floor..
  Post-anesthesia opioid use is measured in milligrams (Morphine Equivalent table) and tracked in the PACU to manage pain. Lower use suggests reasonable pain control; higher use indicates more pain and inadequate control.
Post-Anesthesia Care Unit Stay | Approximately 2-4 hours: From the moment the patient arrives in the Post Anesthesia Care Unit (PACU) until their departure to the floor..
  The Aldrete Score, used in the PACU, rates from 0 to 10 for discharge readiness. Higher scores mean patients' vital signs are stable; lower scores require more recovery time.
Postoperative complications: | Monitoring for PONV, DVT, and cardiac/pulmonary issues occurs at 24, 48, and 72 hours post-admission for observation.
  We are monitoring post-op complications like episodes of postoperative nausea and vomiting (PONV) with the "PONV impact Scale" in the postoperative care unit, the presence of infections, thrombosis (DVT), and pulmonary and heart issues. PONV will be assessed in PACU; a score ≥5 on the PONV Scale is significant.
Post-Surgery Hospital Stay | Post-surgery stay is hospital typically 7-10 days for recovery and complication management. Extended stays may signal recovery delays.
  The period between the end of the surgical procedure and hospital discharge.

SECONDARY OUTCOMES:
Cognitive impairment and delirium | We measure at two point 1) Pre-operative 2) on post operative day one
  The Mini-Cognitive Assessment Instrument (Mini-Cog) Test is a quick screening tool used to identify possible cases of cognitive impairment. It combines a three-item memory test and a clock-drawing task and is typically used in settings where time is a constraint. If a score below three is obtained, it raises concerns about dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Haleh Saadat, Principal Investigator — Integrated Anesthesia Associates, LLC - Fairfield Division

IPD SHARING:
Plan to Share IPD: No
The investigators have decided not to share individual participant data from this study. This decision is based on the need to rigorously protect the privacy and confidentiality of our participants. Although sharing data can be beneficial for broader research purposes, our primary concern is ensuring that personal health information remains secure and private. Additionally, the specific nature of our study data may not easily lend itself to broader application without detailed context, which could be challenging to provide adequately in a data-sharing scenario.

REFERENCES:
- [Background] Parry SM, Puthucheary ZA. The impact of extended bed rest on the musculoskeletal system in the critical care environment. Extrem Physiol Med. 2015 Oct 9;4:16. doi: 10.1186/s13728-015-0036-7. eCollection 2015. PMID 26457181
- [Background] Tagliafico AS, Torri L, Signori A. Treatment of meralgia paresthetica (Lateral Femoral Cutaneous Neuropathy): A meta-analysis of ultrasound-guided injection versus surgery. Eur J Radiol. 2021 Jun;139:109736. doi: 10.1016/j.ejrad.2021.109736. Epub 2021 Apr 26. PMID 33933838
- [Background] Gupta G, Radhakrishna M, Tamblyn I, Tran DQ, Besemann M, Thonnagith A, Elgueta MF, Robitaille ME, Finlayson RJ. A randomized comparison between neurostimulation and ultrasound-guided lateral femoral cutaneous nerve block. US Army Med Dep J. 2017 Jul-Sep;(2-17):33-38. PMID 28853117
- [Background] Neuman MD, Feng R, Carson JL, Gaskins LJ, Dillane D, Sessler DI, Sieber F, Magaziner J, Marcantonio ER, Mehta S, Menio D, Ayad S, Stone T, Papp S, Schwenk ES, Elkassabany N, Marshall M, Jaffe JD, Luke C, Sharma B, Azim S, Hymes RA, Chin KJ, Sheppard R, Perlman B, Sappenfield J, Hauck E, Hoeft MA, Giska M, Ranganath Y, Tedore T, Choi S, Li J, Kwofie MK, Nader A, Sanders RD, Allen BFS, Vlassakov K, Kates S, Fleisher LA, Dattilo J, Tierney A, Stephens-Shields AJ, Ellenberg SS; REGAIN Investigators. Spinal Anesthesia or General Anesthesia for Hip Surgery in Older Adults. N Engl J Med. 2021 Nov 25;385(22):2025-2035. doi: 10.1056/NEJMoa2113514. Epub 2021 Oct 9. PMID 34623788
- [Background] O'Connor MI, Switzer JA. AAOS Clinical Practice Guideline Summary: Management of Hip Fractures in Older Adults. J Am Acad Orthop Surg. 2022 Oct 15;30(20):e1291-e1296. doi: 10.5435/JAAOS-D-22-00125. Epub 2022 Jun 17. PMID 36200817
- [Background] Wan HY, Li SY, Ji W, Yu B, Jiang N. Fascia Iliaca Compartment Block for Perioperative Pain Management of Geriatric Patients with Hip Fractures: A Systematic Review of Randomized Controlled Trials. Pain Res Manag. 2020 Nov 25;2020:8503963. doi: 10.1155/2020/8503963. eCollection 2020. PMID 33294087
- [Background] Cai L, Song Y, Wang Z, She W, Luo X, Song Y. The efficacy of fascia iliaca compartment block for pain control after hip arthroplasty: A meta-analysis. Int J Surg. 2019 Jun;66:89-98. doi: 10.1016/j.ijsu.2018.12.012. Epub 2019 Jan 24. PMID 30685517
- [Background] Brown MT, Brangman SA, Smith NH. Early Identification of Cognitive Impairment: Utility of the Mini-Cog in Non-Clinical Settings. J Appl Gerontol. 2023 Oct;42(10):2139-2147. doi: 10.1177/07334648231175606. Epub 2023 May 24. PMID 37224462
- [Background] Clevenger CK, Schlenger A, Gunter D, Glasgow GB. Cognitive assessment in primary care: Practical recommendations. Nurse Pract. 2023 Jul 1;48(7):26-35. doi: 10.1097/01.NPR.0000000000000067. PMID 37368555
- [Background] American Society of Anesthesiologists. Practice advisory for the management of perioperative hypersensitivity and allergic reactions: an updated report by the American Society of Anesthesiologists Task Force on Perioperative Hypersensitivity and Allergic Reactions. Anesthesiology. 2020;133(1):169-192
- [Background] Iwakiri M, Inoue R, Uchida K. Allergic reactions to propofol in adult patients with egg or soybean allergy: a retrospective cohort study from a large database of a single institute. JA Clin Rep. 2023 Jan 9;9(1):1. doi: 10.1186/s40981-022-00591-8. PMID 36617591
- [Background] Apfelbaum JL, Silverstein JH, Chung FF, Connis RT, Fillmore RB, Hunt SE, Nickinovich DG, Schreiner MS, Silverstein JH, Apfelbaum JL, Barlow JC, Chung FF, Connis RT, Fillmore RB, Hunt SE, Joas TA, Nickinovich DG, Schreiner MS; American Society of Anesthesiologists Task Force on Postanesthetic Care. Practice guidelines for postanesthetic care: an updated report by the American Society of Anesthesiologists Task Force on Postanesthetic Care. Anesthesiology. 2013 Feb;118(2):291-307. doi: 10.1097/ALN.0b013e31827773e9. No abstract available. PMID 23364567
- [Background] Ganesh R, Kebede E, Mueller M, Gilman E, Mauck KF. Perioperative Cardiac Risk Reduction in Noncardiac Surgery. Mayo Clin Proc. 2021 Aug;96(8):2260-2276. doi: 10.1016/j.mayocp.2021.03.014. Epub 2021 Jul 3. PMID 34226028
- [Background] Yajnik M, Kou A, Mudumbai SC, Walters TL, Howard SK, Edward Kim T, Mariano ER. Peripheral nerve blocks are not associated with increased risk of perioperative peripheral nerve injury in a Veterans Affairs inpatient surgical population. Reg Anesth Pain Med. 2019 Jan;44(1):81-85. doi: 10.1136/rapm-2018-000006. PMID 30640657
- [Background] Neal JM, Barrington MJ, Brull R, Hadzic A, Hebl JR, Horlocker TT, Huntoon MA, Kopp SL, Rathmell JP, Watson JC. The Second ASRA Practice Advisory on Neurologic Complications Associated With Regional Anesthesia and Pain Medicine: Executive Summary 2015. Reg Anesth Pain Med. 2015 Sep-Oct;40(5):401-30. doi: 10.1097/AAP.0000000000000286. PMID 26288034
- See also: Hip fractures from American Academy of orthopedic Surgeons (AAOS).Cited 2023 May 21 — https://orthoinfo.aaos.org/en/diseases--conditions/hip-fractures